CLINICAL TRIAL: NCT04481178
Title: A Retrospective Study on Laser Treatment of Nevus of Ota in Thai Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Other Study IDs: si347/2020
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Focus on Laser Treatment of Nevus of Ota in Thai Patients
Keywords: Nevus of Ota, laser treatment, Thai
MeSH Terms: conditions — Nevus of Ota | interventions — Lasers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with nevus of Ota: patients with nevus of Ota who had been treated with laser at Siriraj hospital
  Interventions: Other: Laser (QS, Picosecond laser)

INTERVENTIONS:
Other: Laser (QS, Picosecond laser) — QS-Nd Yag Laser, Picosecond laser

SUMMARY:
A retrospective study on efficacy and complication of laser treatment (Q-switched Nd:YAG and picosecond laser) of nevus of Ota in Thai patients

DETAILED DESCRIPTION:
Nevus of Ota is a benign dermal melanocytic nevus found most commonly in Asians. About 50-60% of all cases have the age of onset at birth or within the first year of life, others appear before puberty. It typically presents as a unilateral mottled blue-gray macules and patches distributed along the first and second branches of trigeminal nerve. Due to its marked hyperpigmentation on the face which does not resolved spontaneously, patients may experience psychosocial disturbances and often seek for treatments. Based on selective photothermolysis theory, Q-switched lasers (ruby 694nm, alexandrite 755nm, Nd:YAG 1064nm) have been used for the treatment of nevus of Ota with a success rate of 95% after 6-8 sessions. Reported complications from the lasers are hypopigmentation(15.3%), hyperpigmentation(2.9%), texture changes (2.9%), and scarring (1.9%). Siriraj Skin Laser Center provides laser treatment for nevus of Ota using mainly Q-switched Nd:YAG laser and Picosecond laser. The study of efficacy and complications of Q-switched Nd:YAG and Picosecond laser in the treatment of Nevus of Ota in Thai patients has never been reported. Therefore, we conduct a retrospective study on efficacy and complication of laser treatment (Q-switched Nd:YAG and picosecond laser) of nevus of Ota in Thai patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Nevus of Ota
* Complete data between January 2008 - December 2018

Exclusion Criteria:

* Incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Nevus of Ota
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of laser treatment in paitients with Nevus of Ota | 2008-2018
  Fading of lesions after treatment by chart review

SECONDARY OUTCOMES:
Complication of laser such as hyperpigmentation, hypopigmentation, and scars | 2008-2018
  Complication of laser such as hyperpigmentation, hypopigmentation, and scars
Relapse rate after laser treatment | 2008-2018
  rate of recurrence after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Achavanuntakul P, Manuskiatti W, Wanitphakdeedecha R, Jantarakolica T. Early Treatment Initiation Improves Outcomes in Nevus of Ota: A 10-Year Retrospective Study. Am J Clin Dermatol. 2022 Jan;23(1):105-114. doi: 10.1007/s40257-021-00637-0. Epub 2021 Oct 24. PMID 34693508